CLINICAL TRIAL: NCT00552448
Title: Use of High Frequency Chest Compression (HFCC) in Pediatric Status Asthmaticus
Brief Title: Use of High Frequency Chest Compression in Pediatric Status Asthmaticus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Continuing review not submitted to IRB within 365 days.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20076812
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Pediatric, Asthma, Acute Exacerbation, Pediatric ICU
Keywords: Pediatric, asthma, pediatric ICU
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Use of the HFCC device in addition to standard therapy for status asthmaticus. The use of HFCC will not affect the therapy received
  Interventions: Device: High Frequency Chest Compression VEST
- 2 (No Intervention): This group will not use the VEST or HFCC. They will just have standard therapy for status asthmaticus. The standard therapy will not be affected if they are in this group.

INTERVENTIONS:
Device: High Frequency Chest Compression VEST — every 6 hours for 20 minutes
  Arms: 1

SUMMARY:
Asthma is a disease resulting in mucus hypersecretion and airways obstruction. This causes difficulty breathing. The High Frequency Chest Compressor (HFCC) is a device that has been shown to decrease respiratory complications in individuals with severe disability who are unable to clear airway secretions. There is a lack of studies using this device in children with asthma. The device has been shown in a study to be safe in children with asthma. The investigators propose that using this device in our pediatric patients hospitalized in the pediatric ICU with asthma will result in decreased pediatric ICU stay. The investigators will also look at asthma severity, total days of hospital stay and chest discomfort while on therapy.

DETAILED DESCRIPTION:
Background: Asthma is the third largest cause of hospitalization in children under 15 years of age. It is a reversible obstructive lung disease caused by airway inflammation and constriction of the airway smooth muscle. Mucus producing glands of the airway become enlarged resulting in overproduction of mucus. All those factors result in airflow obstruction with airtrapping, ventilation/perfusion mismatch and hypoxia. Therapies such as beta-agonists (i.e. albuterol), anti-cholinergics (i.e. atrovent) and steroids are used for an acute asthma attack. Unfortunately, patients may develop status asthmaticus, in which a severe attack does not respond to nebulized bronchodilators, and require intensive care admission.

HFCC is an FDA (1988 under Class II 510K) approved device/modality of chest physiotherapy which has been utilized in patients with mucus hypersecretion, atelectasis and pneumonia. There is a paucity of pediatric studies. A comparative retrospective/prospective data analysis on exacerbations and hospitalizations in medically fragile (profoundly disabled) children using outpatient HFCC showed that use of this therapy reduced days of hospitalization for pulmonary exacerbations. Long term use in quadriplegic children reduced pulmonary secretions, incidence of pneumonia, and number of hospitalizations. In the pediatric cystic fibrosis population, there was improvement of lung function during hospitalization and long term decrease in progression of lung disease. Furthermore, in patients with mild to moderate asthma, there was no decline in lung function with the use of beta agonist and HFCC versus beta agonist alone indicating good tolerance and safety.

Because asthma patients have mucus hypersecretion and this modality has been shown to be effective in other patient populations with mucus hypersecretion, this modality can be used as a means of reducing pulmonary morbidity and thereby allowing the respiratory therapist to allocate his/her time more efficiently.

Purpose:

Assess efficacy of HFCC in PICU population ages 2 to 21 years of age with status asthmaticus

Design: Prospective Randomized non blinded HFCC (administered 4 times a day for 20 minutes) with conventional PICU management of asthma exacerbation vs. conventional PICU management of asthma exacerbation alone. Child would not have any of the standard asthma medications changed or stopped because of this study.

End Points of Interest:

Primary

1) PICU days - Average number of PICU days as researched is about 4.47 days. There may be factors such as non PICU floor availability and PICU rounds that may delay transfer from PICU to the non PICU floor. So the official discharge from PICU will be when the attending PICU physician announces or deems it acceptable for PICU discharge

Secondary

1. Length of hospitalization
2. Pediatric Asthma Severity Score a validated asthma severity score in pediatric population: 1) observed level of respiratory distress 2) accessory muscle use 3) auscultation (degree of wheezing) 4) oxygen saturation 5) respiratory rate Scored observations 0, 1, or 2 and total the observation numbers for a Severity score
3. Discomfort

Patient inclusion 2 to 21 yo (VEST approved for over two yo) Admitted to PICU for status asthmaticus Negative urine pregnancy test prior to initiation of study in those with menses

Patient Exclusion

Absolute contraindication to VEST use:

1. Unstable head or neck injury
2. Active hemorrhage with hemodynamic instability
3. Intracranial pressure > 20 mmHg or those in whom intracranial pressures should be avoided (was a relative contraindication but after discussion moved to absolute)

Presence of anomalies such as:

1. Former premature infant with BPD
2. Congenital bronchogenic or pulmonary anomaly (i.e. CF)
3. Congenital heart disease

ELIGIBILITY:
Inclusion Criteria:

* 2 to 21 yo (VEST approved for over two yo) Admitted to PICU for status asthmaticus Negative urine pregnancy test prior to initiation of study in those with menses

Exclusion Criteria:

* Absolute contraindication to VEST use:

  1. Unstable head or neck injury
  2. Active hemorrhage with hemodynamic instability
  3. Intracranial pressure > 20 mmHg or those in whom intracranial pressures should be avoided (was a relative contraindication but after discussion moved to absolute)

Presence of anomalies such as:

1. Former premature infant with BPD
2. Congenital bronchogenic or pulmonary anomaly (i.e. CF)
3. Congenital heart disease

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaobi C Kanu, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (3):
- United States (3):
  - Stony Brook University Medical Center, Stony Brook, New York
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Texas Tech University Health Sciences Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Status Asthmatics Patients on HFCC Device: Use of the HFCC device in addition to standard therapy for status asthmaticus. The use of HFCC will not affect the therapy received
  High Frequency Chest Compression VEST: every 6 hours for 20 minutes
- Pediatric Status Asthmaticus Patients Not Using HFCC: This group will not use the VEST or HFCC. They will just have standard therapy for status asthmaticus. The standard therapy will not be affected if they are in this group.
Period: Overall Study
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Started | 20 | 16
Completed | 19 | 16
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.95 (3.53) | 6.69 (3.93) | 6.28 (3.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 7 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 9 | 9 | 18
  Caucasian | 9 | 2 | 11
  Hispanic or Latino | 1 | 2 | 3
  Two or more Ethnicity/Races | 1 | 1 | 2
  Ethnicity/Race Unknown | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36
Prior Hospitalizations [Number; unit: participants]
  Yes | 11 | 8 | 19
  None | 8 | 8 | 16
  Unknown | 1 | 0 | 1
Home asthma medication [Number; unit: participants] — Please note that because one subject may be on multiple classes of medication so the numbers will not add up
  participants
    None | 1 | 2 | 3
    Bronchodilator alone | 8 | 7 | 15
    Inhaled steroid | 5 | 3 | 8
    Inhaled steroid-long acting bronchodilator | 4 | 1 | 5
    leukotriene receptor antagonist | 6 | 5 | 11
    Antihistamine | 3 | 2 | 5
    Systemic steroid | 2 | 0 | 2
Modified Pulmonary Index Score (Initial) [Mean (Standard Deviation); unit: units on a scale] — Modified Pulmonary Index Score (MPIS): a validated asthma severity score in pediatric population (Carroll CL et al. A modified pulmonary index score with predictive value for pediatric asthma exacerbations, Ann Allergy Asthma Immunol 2005) Consists of: 1) oxygen saturation on room air 2) accessory muscle use 3) inspiratory to expiratory ratio 4) degree of wheezing 5) heart rate 6) respiratory rate. Scored observations 0, 1, 2 or 3. Total score range 0-18.
  Mild exacerbation total less than 6, moderate exacerbation 6 - 10, severe exacerbation higher than 10
  units on a scale | 5.76 (2.91) | 6.42 (2.91) | 6.03 (2.87)

OUTCOME MEASURES:

1. Primary Outcome: Hours Spent in Pediatric ICU
Description: Length of stay (hours) in Pediatric ICU.
Time Frame: Number of hours from admission to discharge from PICU
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Number analyzed (Participants) | 19 | 16
Hours | 23.71 (8.33) | 23.76 (12.24)

2. Secondary Outcome: Total Days of Hospital Admission
Description: This is limited due to non collection by collaborating centers.
Time Frame: Days
Population: Data not collected
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pediatric Asthma Severity Score (Modified Pulmonary Index Score)
Description: Modified Pulmonary Index Score (MPIS): a validated asthma severity score in pediatric population (Carroll CL et al. A modified pulmonary index score with predictive value for pediatric asthma exacerbations, Ann Allergy Asthma Immunol 2005) Consists of: 1) oxygen saturation on room air 2) accessory muscle use 3) inspiratory to expiratory ratio 4) degree of wheezing 5) heart rate 6) respiratory rate Scored observations 0, 1, 2 or 3. Total score range 0 - 18. Mild exacerbation total less than 6, moderate exacerbation 6 - 10, severe exacerbation higher than 10
Time Frame: Discharge from PICU
Population: Participants with available data
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Number analyzed (Participants) | 18 | 13
units on a scale | 1.88 [0 to 5] | 1.9 [0 to 4]

4. Secondary Outcome: Number of Participants With Chest Discomfort
Time Frame: During PICU admission
Measure: Number; unit: participants
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Number analyzed (Participants) | 20 | 16
participants | 3 | 0

ADVERSE EVENTS:
Arm/Group | Pediatric Status Asthmatics Patients on HFCC Device | Pediatric Status Asthmaticus Patients Not Using HFCC
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 3/20 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Status Asthmatics Patients on HFCC Device (N=20) | Pediatric Status Asthmaticus Patients Not Using HFCC (N=16)
Chest discomfort (anticipated) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Chest discomfort was the only anticipated adverse event - there were no unanticipated adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No